CLINICAL TRIAL: NCT06705374
Title: Central Venous Pressure and Right Atrial Pressure Measurements in Supine, Semi-recumbent and Trendelenburg Position
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Carl Sjödin, PhD student, Vastra Gotaland Region
Other Study IDs: CVP/RAP
Record Dates: First submitted 2024-04-30; First posted 2024-11-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive care is directed towards patients with severe illness or risk of serious outcomes following, for example, surgery. Central venous pressure (CVP) is an important part of the hemodynamic assessment of patients in surgery and the intensive care unit (ICU). CVP is normally measured via a central venous catheter (CVC) inserted through the subclavian or internal jugular vein, with the tip placed at the junction to the right atrium. A pressure tubing is connected to one of the branches of the CVC and then connected to a pressure sensor that sends a digital signal to the monitoring screen where CVP can be read in mmHg. To accurately read CVP, the pressure sensor must be positioned at the level of the right atrium. Different external reference points are used nationally and internationally to locate the correct height for the pressure sensor. This study aims to investigate the most commonly used external reference points for CVP measurement in various body positions compared to CVP measured via a solid state pressure catheter in the right atrium (RAP).

DETAILED DESCRIPTION:
A Millar Mikro-Cath solid state pressure catheter is inserted through one of the medial lines of the CVC and guided in position by the pressure curve and verified in position by ultrasound.

CVP is compared to RAP in supine, semi-recumbent, Trendelenburg and lateral position.

CVP, RAP and arterial pressure is recorded in each session with Biopac Acqnowledge.

In each body position PEEP is raised 5 cmH20 and then lowered 5 cmH20.

Ventilator settings, capillary refill time, perfusion index are collected in each setting and before and after PEEP adjustments.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients in mechanical ventilation with an arterial line and a four or five lumen CVC.

Exclusion Criteria:

* under 18 years of age
* in a dynamic phase of their illness i.e. ongoing treatment of severe circulatory or respiratory failure
* positive end-expiratory pressure (PEEP) >14 cmH20 or intolerance to change of body position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients, in mechanical ventilation, sedated to RASS -4 or -5 in mechanical ventilation with a 4 or 5 line CVC.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in mmHg between Right atrial pressure (RAP) and Central venous pressure (CVP) in supine position | 3 minutes after body position change
  Difference in mmHg between RAP (Millar Micro-Cath) and CVP.
Difference in mmHg between RAP and CVP in semi-recumbent position | 3 minutes after body position change
  Difference in mmHg between RAP (Millar Micro-Cath) and CVP.
Difference in mmHg between RAP and CVP in Trendelenburg position | 3 minutes after body position change
  Difference in mmHg between RAP (Millar Micro-Cath) and CVP.
Difference in mmHg between RAP and CVP in right lateral position | 3 minutes after body position change
  Difference in mmHg between RAP (Millar Micro-Cath) and CVP.
Difference in mmHg between RAP and CVP in left lateral position | 3 minutes after body position change
  Difference in mmHg between RAP (Millar Micro-Cath) and CVP.

SECONDARY OUTCOMES:
Change in hemodynamic parameters after body position change | 3 minutes after body position change
  Change in CVP (mmHg)
Change in hemodynamic parameters after PEEP change | 1 minutes after PEEP change
  Change in RAP (mmHg)
Change in hemodynamic parameters after body position change | 3 minutes after body position change
  Change in arterial pressure (mmHg)
Change in hemodynamic parameters after body position change | 3 minutes after body position change
  Change in perfusion index (%)
Change in hemodynamic parameters after body position change | 3 minutes after body position change
  Change in capillary refill time change (sek)
Change in hemodynamic parameters after body position change | 3 minutes after body position change
  Change in RAP (mmHg)
Change in hemodynamic parameters after PEEP change | 1 minutes after PEEP change
  Change in CVP (mmHg)
Change in hemodynamic parameters after PEEP change | 1 minutes after PEEP change
  Change in arterial pressure (mmHg)
Change in hemodynamic parameters after PEEP change | 1 minutes after PEEP change
  In capillary refill time change (sek)
Change in hemodynamic parameters after PEEP change | 1 minutes after PEEP change
  Change in perfusion index (%)

CONTACTS AND LOCATIONS:
Overall Officials: Lotta Johansson, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All excel data that underlie results in publication
Supporting Information: Study Protocol, SAP, ICF